CLINICAL TRIAL: NCT04345497
Title: A Randomized Controlled Trial to Determine the Effects of a Diabetes-specific Formula on Long-term Glycemic Control and Short-term Glycemic Variability in Individuals With Type 2 Diabetes
Brief Title: Diabetes-Specific Formula on Long Term Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BL46
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Determine the effects of a diabetes-specific formula [1-2 servings per day as a (partial) meal replacement] in addition to standard of care on HbA1c level, in comparison with the standard of care only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diabetes-Specific Formula (Experimental): Diabetes-specific formula 1-2 servings a day and Standard of Care
  Interventions: Other: Diabetes-Specific Formula
- Standard of Care (Other): Standard of Care
  Interventions: Other: Standard Of Care

INTERVENTIONS:
Other: Diabetes-Specific Formula — Diabetes-Specific Formula and Standard of Care
  Arms: Diabetes-Specific Formula
Other: Standard Of Care — Standard of Care
  Arms: Standard of Care

SUMMARY:
The study aims to investigate the effect of a diabetes-specific formula (DSF) used as a (partial) meal replacement on long-term glycemic control and short-term glycemic variability in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
This is a randomized, controlled, parallel study. Eligible participants will be randomly allocated (at 1 :1 ratio) to one of two groups: DSF group or control group.The total expected duration of the study is 97 days.

There are two periods in the study:

i) "Run-in Period" (Study Days -6 to -1): participants will wear the CGMS:Continuous Glucose Monitoring System (FreeStyle Libre Pro) and will be asked to follow and track their diet and physical activity on a daily basis.

ii) "Intervention Period" (Study Days 0 to 90): participants will be randomized into one of the two groups (n = 125 per group): DSF group or control group.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants (≥ 21 and ≤ 65 years of age)
2. Has type 2 diabetes as evidenced with oral anti-diabetic drug(s) at constant dose for at least two months prior to the study and is able to maintain number of medications, type and dose throughout the duration of the study
3. BMI ≥ 23 and < 35.0 kg/m2
4. Weight is stable (has maintained current body weight within 3 kg) for the two months prior to the Baseline Visit
5. Either a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to the Baseline Visit. A urine pregnancy test is required for all female participants unless she is not of childbearing potential, defined as postmenopausal for at least one year prior to the Baseline Visit or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
6. If the female is of childbearing potential, she is practicing one of the following methods of birth control and will continue through the duration of the study:

   1. Condoms, sponge, diaphragm or intrauterine device;
   2. Oral or parenteral contraceptives for 3 months prior to Baseline Visit;
   3. Vasectomized partner;
   4. Total abstinence from sexual intercourse
7. If on a chronic medication such as an anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, the medication number, type and dose were constant for at least two months prior to the Baseline Visit and will continue through the duration of the study
8. Willingness to follow the protocol as described, including consumption of study product per the protocol and completing any forms/questionnaires needed throughout the study
9. At least a two-week washout period is needed between the completion of a previous research study that required ingestion of any study food or drug and their start in the current study
10. The participant is willing to refrain from taking non-study diabetes-specific formulas over the entire course of the study

Exclusion Criteria:

1. Screening HbA1c level <7% or ≥ 10%
2. Use of exogenous insulin for glucose control
3. Confirmed type 1 diabetes and/or had a history of diabetic ketoacidosis
4. Current infection (requiring medication), inpatient surgery or received systemic corticosteroid treatment [except for inhaled (includes nasal), topical, and ophthalmic steroids] in the last 3 months; or received antibiotics in the last 3 weeks
5. Active malignancy within the last 5 years
6. A significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure
7. End-stage organ failure (such as end-stage renal disease) or is post-organ transplant
8. Current or history of renal disease or on dialysis or severe gastroparesis
9. Current hepatic disease
10. Has had bariatric surgery including gastric balloon; the history of gastrointestinal disease (e.g., Crohn's, colitis, celiac) or intestinal surgery that can interfere with consumption or digestion or absorption of study product
11. A chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV
12. Has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures in the opinion of the principal investigator or study physician
13. Taking any herbals, dietary supplements, or medications during the past four weeks prior to Baseline Visit that could profoundly affect (in the opinion of the primary investigator) blood glucose or appetite (e.g. orlistat, contrive, qsymia, belviq, incretins, cannabis, glucocorticoids, nicotinic acid, etc.) per healthcare professional's opinion
14. Using diabetes-specific formula(s), (e.g. Glucerna, Nestle Nutren Diabetes, Kalbe Diabetasol, Appeton Nutrition Wellness 60+ Diabetic, ForSure, Penta Sure DM, Resurge DM, Diben, Diasip, etc.) defined as more than one eating occasion per week within the past 3 months (those users who have stopped using such products for more than 3 months may not be excluded)
15. Clotting or bleeding disorders (the use of Plavix® or a similar anticoagulant drug with no reported difficulty during blood draws will be allowed)
16. Has blood or blood-related diseases (e.g. hemophilia, thalassemia, sickle cell disease, hereditary spherocytosis, glucose-6-phosphate dehydrogenase deficiency)
17. Received a blood transfusion within the last 3 weeks
18. Allergic or intolerant to any ingredient found in the test meals
19. Participates in another study that has not been approved as a concomitant study by Abbott Nutrition
20. The participant has skin lesions hyperhidrosis, eczema, psoriasis, scarring, tattoos, redness, infection or edema at the application sites that in the opinion of the study investigator or study physician could interfere with device placement or the accuracy of interstitial glucose measurements.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
HbA1c Level | Study Days 0, 45 and 90
  Change in HbA1c level from Day 0 to Day 90

SECONDARY OUTCOMES:
Glycemic Excursion | Study Day 1 to Day 7
  Mean Amplitude of Glycemic Excursions (MAGE)
Glucose | Study Day 1 to Day 7
  Mean and coefficient of variation (CV) of glucose during the intervention phase
Time of glucose level | Study Day 1 to Day 7
  Time of glucose level in target, below and above range per day during intervention phase
Hypoglycemic Episodes | Study Day 1 to Day 7
  Number of hypoglycemic episodes per day during the intervention phase
Hyperglycemic Episodes | Study Day 1 to Day 7
  Number of hyperglycemic episodes per day during the intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Siew Ling Tey, Ph.D., Study Chair — Abbott Nutrition
Locations (5):
- Malaysia (3):
  - International Medical University, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
  - Klinik Kesihatan Seremban, Seremban
- Thailand (2):
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok